CLINICAL TRIAL: NCT04659044
Title: A Phase 2 Trial of the Combination of Polatuzumab Vedotin, Venetoclax and Rituximab and Hyaluronidase Human for Relapsed and Refractory Mantle Cell Lymphoma
Brief Title: Polatuzumab Vedotin, Venetoclax, and Rituximab and Hyaluronidase Human for the Treatment of Relapsed or Refractory Mantle Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial closed due to low accrual rate
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-LY-1806; NCI-2020-08188 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-LY-1806 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2020-11-19; First posted 2020-12-09 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3a Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Grade 1 Follicular Lymphoma; Refractory Grade 2 Follicular Lymphoma; Refractory Grade 3a Follicular Lymphoma; Refractory Mantle Cell Lymphoma; Refractory Marginal Zone Lymphoma; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — polatuzumab vedotin; Rituximab; CT-P10; Hyaluronoglucosaminidase; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (rituximab, polatuzumab vedotin, venetoclax) (Experimental): INDUCTION: Patients receive rituximab IV on day 1 of cycle 1 and rituximab and hyaluronidase human SC over 5 minutes on day 1 of cycles 2-6. Patients also receive polatuzumab vedotin IV over 30-90 minutes on day 1 and venetoclax PO daily on days 1-21. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive venetoclax PO daily on days 1-21 and rituximab and hyaluronidase human SC over 5 minutes every 60 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Polatuzumab Vedotin; Biological: Rituximab; Biological: Rituximab and Hyaluronidase Human; Drug: Venetoclax

INTERVENTIONS:
Drug: Polatuzumab Vedotin — Given IV
  Other Names: ADC DCDS4501A; Antibody-Drug Conjugate DCDS4501A; DCDS4501A; FCU 2711; polatuzumab vedotin-piiq; Polivy; RG7596; Ro 5541077-000
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Riabni; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; rituximab-abbs; Rituximab-arrx; Rituximab-pvvr; RTXM83; Ruxience; Truxima
Biological: Rituximab and Hyaluronidase Human — Given SC
  Other Names: Rituxan Hycela; Rituximab Plus Hyaluronidase; Rituximab/Hyaluronidase; Rituximab/Hyaluronidase Human
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies the effect of polatuzumab vedotin, venetoclax, and rituximab and hyaluronidase human in treating patients with mantle cell lymphoma that has come back (relapsed) or does not respond to treatment (refractory). Polatuzumab vedotin is a monoclonal antibody, polatuzumab, linked to a toxic agent called vedotin. Polatuzumab attaches to CD79B positive cancer cells in a targeted way and delivers vedotin to kill them. Venetoclax may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cell growth. Rituximab hyaluronidase is a combination of rituximab and hyaluronidase. Rituximab binds to a molecule called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. This may help the immune system kill cancer cells. Hyaluronidase allows rituximab to be given by injection under the skin. Giving rituximab and hyaluronidase by injection under the skin is faster than giving rituximab alone by infusion into the blood. Giving polatuzumab vedotin, venetoclax, and rituximab and hyaluronidase human may work better than standard therapy in treating patients with mantle cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the end of induction (EOI) complete response rate (CR) for treatment with the regimen of rituximab and hyaluronidase human + polatuzumab vedotin + venetoclax (RSc + Pola + Ven) in relapsed/refractory mantle cell lymphoma (MCL).

SECONDARY OBJECTIVES:

I. To evaluate the EOI overall response rate (ORR) for the combination of RSc + Pola + Ven in relapsed/refractory MCL.

II. To evaluate the best response (CR, partial response [PR]) in patients who continue on to maintenance therapy and evaluate the improvement in the depth of response.

III. To evaluate the progression free survival (PFS) and overall survival (OS) for the combination of RSc + Pola + Ven) in relapsed/ refractory MCL.

IV. To compare the ORR, CR, PFS, and OS in ibrutinib refractory compared to ibrutinib naive patients.

V. To evaluate regimen-related toxicity for patients treated with RSc + Pola + Ven.

CORRELATIVE RESEARCH OBJECTIVES:

I. To evaluate changes in minimal residual disease (MRD) status in both responding and non-responding patients at EOI and end of maintenance and compared to baseline as well as correlate MRD status with PFS and OS.

II. To evaluate changes in systemic immune profiles and T cell activation induced by treatment with RSc + Pola + Ven.

III. To evaluate the prognostic importance of high risk cytogenetic alterations, and other risk stratification scores in patients with relapsed/refractory MCL receiving RSc + Pola + Ven.

IV. To evaluate features of the tumor microenvironment in patients with relapsed/refractory MCL receiving RSc +Pola+Ven.

V. To evaluate molecular features associated with response in PDX models from patients with relapsed/refractory MCL receiving RSc +Pola+Ven.

OUTLINE:

INDUCTION: Patients receive rituximab intravenously (IV) on day 1 of cycle 1 and rituximab and hyaluronidase human subcutaneously (SC) over 5 minutes on day 1 of cycles 2-6. Patients also receive polatuzumab vedotin IV over 30-90 minutes on day 1 and venetoclax orally (PO) daily on days 1-21. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive venetoclax PO daily on days 1-21 and rituximab and hyaluronidase human SC over 5 minutes every 60 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 90 days for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Pathologically confirmed relapsed or primary refractory mantle cell lymphoma with concurrent or prior tissue sample immunohistochemistry (IHC) positive for cyclin D1 or that is positive for fluorescence in situ hybridization (FISH) or cytogenetics for t(11;14)

  * NOTE: Safety Portion only: MCL or indolent B cell non-Hodgkin lymphoma (NHL), follicular lymphoma (FL) (grades I-IIIa), marginal-zone lymphoma (MZL) or small lymphocytic lymphoma (SLL) stratified as low risk for tumor lysis syndrome (TLS), relapsed or progressed after at least two lines of therapy, or one line of a BTK inhibitor containing therapy, or Autologous Stem Cell Transplant (AutoSCT). No limit to prior lines of therapy
  * NOTE: Expansion Portion only: MCL relapsed or progressed after at least two lines of therapy, or one line of a BTK inhibitor containing therapy, or Autologous Stem Cell Transplant (AutoSCT). No limit to number of prior therapies. May have received prior BTK inhibitor therapy
* Measurable disease as defined with at least one lesion measuring >= 1 x 1.5 cm by positron emission tomography (PET)-computed tomography (CT) using Lugano criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1000/mm^3 (obtained =< 14 days prior to registration)
* Platelet count >= 75,000/mm^3 (obtained =< 14 days prior to registration)
* Hemoglobin >= 9.0 g/dL (obtained =< 14 days prior to registration)
* International normalized ratio =< 1.5 x upper limit of normal (ULN) for patients not receiving therapeutic anticoagulation (obtained =< 14 days prior to registration)
* Partial thromboplastin time (PTT) or activated PTT (aPTT) =< 1.5 x upper limit of normal (ULN) (obtained =< 14 days prior to registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN (obtained =< 14 days prior to registration)
* Total bilirubin < 1.5 x ULN (or =< 3 x ULN for patients with documented Gilbert syndrome) (obtained =< 14 days prior to registration)
* Calculated creatinine (Cr) clearance >= 45 ml/min using the modified Cockcroft-Gault formula (obtained =< 14 days prior to registration)
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only

  * NOTE: A female of childbearing potential is a sexually mature female who:

    * Has not undergone a hysterectomy or bilateral oophorectomy; or
    * Has not been naturally postmenopausal for at least 12 consecutive months (i.e. has had menses at any time in the preceding 12 consecutive months)
* Able to provide informed written consent, and ability to comply with study related procedures
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* Willing to provide tissue samples for mandatory correlative research
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 30 days after the last dose of venetoclax or 18 months after the last dose of rituximab and hyaluronidase human, whichever is longer. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

  * With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 6 months after the last dose. Men must refrain from donating sperm during this same period.
  * With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 6 months after the last dose to avoid exposing the embryo

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational or chemotherapeutic agent which would be considered as a treatment for the primary neoplasm
* Known CD20-negative status at relapse or progression
* Prior allogeneic SCT
* Completion of autologous SCT =< 100 days prior to registration
* Treatment with radioimmunoconjugate =< 12 weeks prior to registration
* Monoclonal antibody or antibody-drug conjugate (ADC) therapy within 5 half-lives or 4 weeks prior to registration, whichever is longer
* Radiotherapy, chemotherapy, hormonal therapy, or targeted small-molecule therapy within 2 weeks prior to registration (with the exception of ibrutinib to prevent tumor flare, patients taking ibrutinib who are progressing must discontinue ibrutinib 2 half-lives or 2 days prior to initiating protocol therapy)
* Clinically significant toxicity (other than alopecia) from prior therapy that has not resolved to grade =< 2 (per National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v]5.0) prior to registration
* Current grade > 1 peripheral neuropathy
* Any history of central nervous system (CNS) lymphoma or leptomeningeal infiltration
* Treatment with systemic corticosteroids > 20 mg/day prednisone or equivalent Patients who are receiving corticosteroids =< 20 mg/day, prednisone or equivalent, for non-lymphoma treatment reasons must be documented to be on a stable dose for >= 4 weeks prior to registration. If corticosteroid treatment is urgently required for lymphoma symptom control prior to the start of study treatment, up to 100 mg/day of prednisone or equivalent can be given for a maximum of 5 days, but all tumor assessments must be completed prior to start of corticosteroid treatment
* History of severe allergic or anaphylactic reaction or known sensitivity to humanized or murine monoclonal antibodies rituximab, polatuzumab vedotin, or venetoclax
* Active bacterial, viral, fungal, or other infection
* Requirement for warfarin treatment (because of potential drug-drug interactions [DDIs] that may increase the exposure of warfarin)
* Treatment with the following agents =< 7 days prior to registration

  * Strong and moderate CYP3A inhibitors such as fluconazole, ketoconazole, and clarithromycin
  * Strong and moderate CYP3A inducers such as rifampin and carbamazepine. If subject is taking proton pump inhibitors, subject is willing to avoid co-administration and stagger venetoclax dosing
* Consumption of grapefruit, grapefruit products, Seville oranges (including marmalade that contains Seville oranges), or star fruit =< 3 days prior to registration
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Active hepatitis B or hepatitis C infection

  * NOTE: Patients who have been successfully treated and cleared their virus as evidenced by a negative hepatitis (Hep) B or Hep C polymerase chain reaction (PCR) are eligible
* Known history of human immunodeficiency virus (HIV) positive status or known infection with human T-cell leukemia virus 1. For patients with unknown HIV status, HIV testing will be performed at screening
* History of PML (progressive multifocal leukoencephalopathy)
* Vaccination with a live virus vaccine =< 28 days prior to registration
* History of other malignancy that could affect compliance with the protocol or interpretation of results, with the exception of the following: curatively treated carcinoma in situ of the cervix, good-prognosis ductal carcinoma in situ of the breast, basal- or squamous-cell skin cancer, stage I melanoma, or low-grade, early-stage localized prostate cancer
* Any previously treated malignancy that has been in remission without treatment for =< 3 years prior to registration
* Evidence of any significant, uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease (such as New York Heart Association class III or IV cardiac disease, myocardial infarction within the previous 6 months, unstable arrhythmia, or unstable angina) or significant pulmonary disease (such as obstructive pulmonary disease or history of bronchospasm)
* Major surgical procedure other than for diagnosis =< 28 days prior to day 1 of cycle 1, or anticipation of a major surgical procedure during the course of the study
* Inability or unwillingness to swallow pills
* History of malabsorption syndrome or other condition that would interfere with enteral absorption
* History of inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis) or active bowel inflammation (e.g., diverticulitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine S Diefenbach, Principal Investigator — Academic and Community Cancer Research United
Locations (5):
- United States (5):
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Rituximab, Polatuzumab Vedotin, Venetoclax): INDUCTION: Patients receive rituximab IV on day 1 of cycle 1 and rituximab and hyaluronidase human SC over 5 minutes on day 1 of cycles 2-6. Patients also receive polatuzumab vedotin IV over 30-90 minutes on day 1 and venetoclax PO daily on days 1-21. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive venetoclax PO daily on days 1-21 and rituximab and hyaluronidase human SC over 5 minutes every 60 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Polatuzumab Vedotin: Given IV
  Rituximab: Given IV
  Rituximab and Hyaluronidase Human: Given SC
  Venetoclax: Given PO
Period: Induction
Arm/Group | Treatment (Rituximab, Polatuzumab Vedotin, Venetoclax)
Started | 3
Completed | 0
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Adverse Event | 2
Period: Maintenance Therapy
Arm/Group | Treatment (Rituximab, Polatuzumab Vedotin, Venetoclax)
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Rituximab, Polatuzumab Vedotin, Venetoclax)
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (19.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 3
ECOG Performance Status [Count of Participants; unit: Participants] — 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    <=1 | 2
    >=2 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing a Complete Response (CR)
Description: Objective status of CR measured by positron emission tomography (PET)-computed tomography (CT) scans according to Lugano 2014.
Time Frame: 3 months
Population: Only patients that had at least one post-baseline disease assessment were included in analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Rituximab, Polatuzumab Vedotin, Venetoclax)
Number analyzed (Participants) | 2
Participants | 0

2. Secondary Outcome: Overall Response Rate (ORR)
Description: The ORR at the end of induction will be estimated by the total number of patients who achieve a complete response (CR) or partial response (PR) by PET-CT scans according to Lugano 2014 divided by the total number of evaluable patients. The ORR between ibrutinib-naive and ibrutinib-pretreated patients will be compared using Fisher's exact test.
Time Frame: 3 months
Population: Only patients that had at least one post-baseline disease assessment were included in analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Rituximab, Polatuzumab Vedotin, Venetoclax)
Number analyzed (Participants) | 2
Participants | 0

3. Secondary Outcome: Best Response Rate to Maintenance Therapy
Description: CR, PR, and stable disease (SD) rates for patients who continue to maintenance will be estimated by number of patients who continue on maintenance therapy and achieve CR, PR or SD, respectively, at the end of maintenance divided by the total number of evaluable patients who continue to maintenance.
Time Frame: At the end of maintenance therapy
Population: No patients were on study long enough to receive maintenance therapy.
Arm/Group | Treatment (Rituximab, Polatuzumab Vedotin, Venetoclax)
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival (PFS)
Description: The distribution of PFS will be estimated using the method of Kaplan-Meier. The PFS between ibrutinib-naive and ibrutinib-pretreated patients will be compared using log-rank test.
Time Frame: 10 months
Population: Only patients that had at least one post-baseline disease assessment were included in analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Rituximab, Polatuzumab Vedotin, Venetoclax)
Number analyzed (Participants) | 2
months | 5.5 [1.1 to NA] — The upper limit of the confidence interval cannot be estimated due to a low number of events.

5. Secondary Outcome: Overall Survival (OS)
Description: The distribution of OS will be estimated using the method of Kaplan-Meier. The OS between ibrutinib-naive and ibrutinib-pretreated patients will be compared using log-rank test.
Time Frame: 15 months
Population: Only patients that had at least one post-baseline disease assessment were included in analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Rituximab, Polatuzumab Vedotin, Venetoclax)
Number analyzed (Participants) | 2
months | NA [1.1 to NA] — The median survival time and upper limit of the confidence interval cannot be estimated due to a low number of events.

6. Secondary Outcome: Count of Patients Experiencing Grade 3+ Adverse Events (AEs)
Description: All AEs occurring on or after first study treatment will be summarized by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 grade.
Time Frame: 15 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Rituximab, Polatuzumab Vedotin, Venetoclax)
Number analyzed (Participants) | 3
Participants | 3

7. Other Pre Specified Outcome: Minimal Residual Disease (MRD) Analysis
Description: MRD status for both responders and non-responders at each time point will be reported descriptively, and explored for correlation with clinical factors and patient outcomes such as PFS and OS.
Time Frame: Up to the end of maintenance therapy
Reporting Status: Not Posted

8. Other Pre Specified Outcome: T Cell and Cytokine Subset Analysis
Description: Systemic immune profiles and T cell activation will be investigated using multi-parameter flow cytometry, and cytokine analysis in the peripheral blood of patients.
Time Frame: Up to the end of maintenance therapy
Reporting Status: Not Posted

9. Other Pre Specified Outcome: High Risk Cytogenetic Alterations
Description: Will be summarized using frequency and percentages.
Time Frame: Up to the end of maintenance therapy
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Risk Stratification Scores
Description: Will be summarized using frequency and percentages.
Time Frame: Up to the end of maintenance therapy
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Treatment (Rituximab, Polatuzumab Vedotin, Venetoclax)
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Rituximab, Polatuzumab Vedotin, Venetoclax) (N=3)
Neutrophil count decreased (Investigations) | 1 (2)
White blood cell decreased (Investigations) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Disease Progression (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Rituximab, Polatuzumab Vedotin, Venetoclax) (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (10)
Anemia (Blood and lymphatic system disorders) | 2 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (8)
Blood lactate dehydrogenase increased (Investigations) | 2 (2)
Cholesterol high (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
GGT increased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (4)
Hypotension (Vascular disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (10)
Malaise (General disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (3)
Pain (General disorders) | 1 (3)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Platelet count decreased (Investigations) | 2 (3)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 2 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT04659044/Prot_SAP_000.pdf